CLINICAL TRIAL: NCT00835601
Title: An Integrated Musculoskeletal Countermeasure Battery for Long-Duration Lunar Missions
Brief Title: Resistive/Cardiovascular Training Study
Acronym: CCD
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Thomas.Lang, PhD/Professor in Residence, UCSF
Other Study IDs: CCD Training Study; NSBRI BL-01301
Record Dates: First submitted 2009-01-29; First posted 2009-02-03 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a training study in healthy volunteers to characterize gains in lower-body resistive strength and cardiovascular capacity with exercise on a Combined Countermeasure Device (CCD) we have developed for the National Space Biomedical Research Institute. The CCD is a single platform which contains interchangeable modules for cardiovascular stepping exercises and lower body resistive exercises including squats, heel raises, abductor and adductor exercises and knee extension and flexion. The platform has the capability to tilt, yaw and pitch, and to translate in three dimensions in order to challenge the neurovestibular system. The underlying goal of the project is to provide a compact and efficient exercise modality that will prevent deterioration of the cardiovascular and musculoskeletal systems, and the neurovestibular system, in long-duration spaceflights. The goal of the current study is simply to test the hypothesis that in healthy volunteers, the exercise prescription proposed for the device will improve strength and VO2 max. Subjects are tested for lower body resistive strength and V02max at baseline, then are trained for 12 weeks, and tested again at followup to test for a change. 36 subjects, allowing for a 20% attrition rate, allows sufficient power to detect 95% percent confidence intervals in the changes in the strength and V02max measures of roughly 10-20%. If we observe gains in these indices which are similar to those reported in the literature for simultaneous cardiovascular and resistive strength protocols, then we believe that there is sufficient evidence to test CCD in a bedrest model of long-duration spaceflight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 25-55 years old
* Do not exercise on a regular basis

Exclusion Criteria:

Have not been diagnosed with hypertension, diabetes, high cholesterol, cardiovascular disease or asthma and other pulmonary disorders

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women 25-55 years of age who are not exercisers
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
VO2max | 6-12 weeks
Leg Press Strength | 6-12 weeks